CLINICAL TRIAL: NCT06018883
Title: Vitamin C to Chemotherapy Related Anemia in Pancreatic Cancer
Acronym: PTCA199-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTCA199-3
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: ascorbate; anemia; quality of life; chemotherapy
MeSH Terms: conditions — Anemia | interventions — Ascorbic Acid; Taxes; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbate (Experimental): nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks. Vitamin C 900 mg/day, three times a day, orally.
  Interventions: Drug: Ascorbate; Drug: Nab paclitaxel; Drug: Gemcitabine
- Control (Other): nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbate — Vitamin C 900 mg/day, three times a day, orally.
  Other Names: Vitamin C
  Arms: Ascorbate
Drug: Nab paclitaxel — Nab-paclitaxel (120 mg per square meter of body-surface area) on days 1, 8, and 15 every 4 weeks
  Other Names: Nab-paclitaxel
Drug: Gemcitabine — Gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks
  Other Names: Gemcitabine Hydrochloride

SUMMARY:
The purpose of this study is to evaluate the efficacy of low-dose vitamin C on improving the quality of life for metastatic pancreatic cancer patients receiving gemcitabine and nab-paclitaxel chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. The Metastatic PAncreatic Cancer Trial (MPACT) has confirmed the efficacy of gemcitabine combined with nab-paclitaxel as the first-line treatment to metastatic pancreatic cancer. However, the side-effects related to gemcitabine combined with nab-paclitaxel including anemia, hand/foot numbness, fatigue, nausea, and malnutrition have impaired the tolerability of the regimen.

Vitamin C, also called ascorbate, is an essential nutrient for the human body. It modulates metabolism, immune reaction, collagen synthesis, and iron absorption. Some studies have shown that high-dose intravenous Vitamin C may be effective against various types of cancer. Meanwhile, medium or low dose of Vitamin C may enhance the tolerability of chemotherapy by increasing iron absorption, improving anemia, alleviating pain and hand/foot numbness, and thus improving quality of life for patients with pancreatic cancer.

The purpose of this study is to evaluate the efficacy of low-dose vitamin C on improving the quality of life for metastatic pancreatic cancer patients receiving gemcitabine and nab-paclitaxel chemotherapy. One hundred patients will be randomly assigned to the experimental group (gemcitabine combined with nab-paclitaxel, Vitamin C) or the control group (gemcitabine combined with nab-paclitaxel). Rate of anemia, rate of hand/foot numbness, severity of pain, quality of life, and overall survival are measured every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
* Adequate organ performance based on laboratory blood tests.
* Presence of at least of one measurable lesion in agreement to Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
* Hemoglobin (Hgb) ≥ 8 g/dL.
* The expected survival ≥ 3 months.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients who have received any form of anti-tumor therapy.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Pregnant or nursing women.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results, including active opportunistic infections or advanced (severe) infections, and diabetes that cannot be controlled after adequate clinical anti-hyperglycemia treatment according to guidelines, uncontrollable hypertension, cardiovascular disease (Class III or IV heart failure as defined by the New York Heart Association classification, congestive heart failure (CHF), myocardial infarction in the past 6 months , unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc).
* Renal insufficiency or dialysis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, nab-paclitaxel, or other agents used in the study.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
* Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Rate of anemia | At the end of Cycle 1 (each cycle is 28 days)
  Rate of anemia after every cycle of chemotherapy

SECONDARY OUTCOMES:
Rate of grade 3 neuropathy | At the end of Cycle 1 (each cycle is 28 days)
  Rate of grade 3 neuropathy after every cycle of chemotherapy
Change of numeric rating scale (NRS) | At the end of Cycle 1 (each cycle is 28 days)
  Change of NRS and the administration of analgesic drugs after every cycle of chemotherapy. The range of NRS scale is 0-10 and higher scores mean a worse outcome.
Quality of life (QOL) | At the end of Cycle 1 (each cycle is 28 days)
  Change of QOL after every cycle of chemotherapy assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Overall survival (OS) | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magri A, Germano G, Lorenzato A, Lamba S, Chila R, Montone M, Amodio V, Ceruti T, Sassi F, Arena S, Abrignani S, D'Incalci M, Zucchetti M, Di Nicolantonio F, Bardelli A. High-dose vitamin C enhances cancer immunotherapy. Sci Transl Med. 2020 Feb 26;12(532):eaay8707. doi: 10.1126/scitranslmed.aay8707. PMID 32102933
- [Background] Drisko JA, Serrano OK, Spruce LR, Chen Q, Levine M. Treatment of pancreatic cancer with intravenous vitamin C: a case report. Anticancer Drugs. 2018 Apr;29(4):373-379. doi: 10.1097/CAD.0000000000000603. PMID 29438178
- [Background] Cieslak JA, Cullen JJ. Treatment of Pancreatic Cancer with Pharmacological Ascorbate. Curr Pharm Biotechnol. 2015;16(9):759-70. doi: 10.2174/138920101609150715135921. PMID 26201606
- [Derived] Wang X, Zhu X, Liu Y, Liu H, Xiao Z, Luo G. Efficacy of vitamin C on chemotherapy-related anemia in pancreatic cancer: study protocol for a randomized controlled trial. Trials. 2024 Jul 29;25(1):512. doi: 10.1186/s13063-024-08345-w. PMID 39075587